CLINICAL TRIAL: NCT07328581
Title: Phase I, IIa, Single-Arm, Study of BCMA-CD19-IL-15/IL15sushi cCAR T for the Treatment of Refractory Systemic Lupus Erythematosus, With or Without Lupus Nephritis
Brief Title: BCMA-CD19 cCAR T for the Treatment of Refractory Lupus
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: iCell Gene Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICG318-001
Record Dates: First submitted 2025-10-17; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus (SLE); Lupus Nephritis (LN)
Keywords: Lupus; autoimmune disease; CAR-T Cell; Refractory disease; CD19; BCMA; Lupus Nephritis (LN); Systemic Lupus Erythrematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis; Autoimmune Diseases; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Biologic drug infusion
  Interventions: Biological: ICG318, BCMA-CD19-IL-15/IL-15 sushi Compound CAR T following cyclophosphamide-only lymphodepletion

INTERVENTIONS:
Biological: ICG318, BCMA-CD19-IL-15/IL-15 sushi Compound CAR T following cyclophosphamide-only lymphodepletion — Anti-BCMA, Anti-CD19 Compound CAR-T Cells

SUMMARY:
This is a Phase I, IIa, Single-Arm, interventional, open label, treatment study to evaluate the safety and tolerability of BCMA-CD19-IL-15/IL15sushi cCAR T cells in patients with relapsed and/or refractory SLE, with or without Lupus Nephritis.

DETAILED DESCRIPTION:
Systemic Lupus Erythematosus (SLE) is a multisystem, chronic autoimmune disease that may impact multiple organs including the joints, skin, kidney, heart, brain and lungs, with severity ranging from mild to life-threatening. Lupus Nephritis (LN) is the most prevalent and severe form of SLE with high morbidity and mortality and persistent relapses despite current therapies.

SLE, with or without LN is driven largely by pathogenic autoantibodies produced by CD19 expressing B cells and BCMA expressing plasma cells, including long-lived plasma cells.

ICG318, the investigational agent in this clinical trial is an armored, compound chimeric antigen receptor (CAR) composed of two independently functioning CARs that simultaneously target the B-cell CD19 surface antigen and the plasma cell/ long lived plasma cell BCMA surface antigen.

This study is being conducted to evaluate the safety and efficacy of ICG318 in SLE patients with or without LN, who have not shown adequate clinical response to prior therapies.

A single dose of ICG318 following a cyclophosphamide-only lymphodepletion regimen will be evaluated.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age 16-70 years at the time of signing the informed consent
2. Have a diagnosis of SLE by EULAR/ACR 2019 criteria for ≥6 months.
3. Have at least one of an antinuclear antibody, anti-double-stranded deoxyribonucleic acid (dsDNA), or elevated anti-Smith (Sm) antibody
4. Inadequate response to 2 prior standard of care therapies, used for at least three months
5. SLE Disease Activity Index 2000 (SLEDAI-2K) score of ≥7 at Screening
6. For LN cohort participants. Kidney biopsy result within 6 months prior to Screening indicating Class III or IV (alone or in combination with Class V)6.

Key Exclusion Criteria:

1. Any acute, severe lupus related flare that needs immediate treatment
2. History of antiphospholipid syndrome with thromboembolic event within 12 months
3. History or current diagnosis of any disease, condition or treatment that may confound clinical assessments in the study.
4. Has drug-induced SLE.
5. History of prior CAR-T therapy.
6. History of bone marrow/hematopoietic stem cell or solid organ transplant or planned receipt during the study period.
7. Recent serious or ongoing infection, or risk for serious infection, or acute or chronic infection
8. Receipt of a live/live-attenuated vaccine other than BCG within 8 weeks
9. History within the past year or current clinically significant central nervous system disease, including but not limited to cerebrovascular accident, seizures, severe brain injury, dementia, Parkinson's disease, cerebellar disease, or multiple sclerosis
10. Impaired cardiac function or clinically significant cardiac disease
11. End stage renal disease or severe liver disease
12. Breastfeeding/lactating or pregnant women or women who intend to become pregnant at any time during the study.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events after ICG318 infusion | Starting day 0 and up to 1 year after ICG318 infusion.
  Number of participants with Adverse Events (AEs), Serious Adverse Events (SAEs), Treatment Emergent Adverse Events (TEAEs), Adverse Events of Special Interest (AESI), and Dose Limiting Toxicities (DLTs).
DORIS remission rate | Starting day 0 and assessed at 6 months, and 1 year after ICG318 infusion.
  DORIS remission defined as no circulating autoantibodies (e.g. dsDNA, Smith etc.) detected, no SLE medications, and SLEDAI-2K score of 0-1 (down from severe 7-10).

SECONDARY OUTCOMES:
Determine the recommended phase 2 dose (RP2D) regimen. | Starting day 0 and assessed 1 year after ICG318 infusion.
  The protocol is based on cohort schema with dose escalation from 0.5x10^6/kg to 4x10^6/kg.
Cmax | Assessed as per schedule of events up to 1 year after ICG318 infusion.
  Maximum serum concentration of ICG318.
Tmax | Assessed as per schedule of events up to 1 year after ICG318 infusion.
  Time to maximum serum concentration of ICG318.
T1/2 | Assessed as per schedule of events up to 1 year after ICG318 infusion.
  Half-life of ICG318 serum concentration.
AUC | Assessed as per schedule of events up to 1 year after ICG318 infusion.
  Plasma ICG318 concentration versus time. Total systemic exposure to ICG318 over time.
Rate of B cell elimination and naïve B-Cell recovery | Assessed as per schedule of events up to 1 year after ICG318 infusion.
  B cell subsets will be assessed by flow cytometry panels and B-Cell receptor sequencing.
Recovery of immunoglobulins | Assessed as per schedule of events up to 1 year after ICG318 infusion.
  Immunoglobulins IgG, IgM and IgA levels.
SLE Autoantibody levels | Assessed as per schedule of events up to 1 year after ICG318 infusion.
  Changes in levels of SLE specific autoantibodies (e.g. dsDNA, Smith etc.)
Number of patients achieving DORIS remission, LLDAS, Complete or Partial Renal Response (in LN patients) | Starting day 0 and assessed at 6 months, and 1 year after ICG318 infusion.
  As per the DORIS and SLEDAI-2K remission criteria.
Renal histology | The first biopsy will be obtained prior to ICG318 infusion. Next biopsy will be assessed up to 6 months to 1 year after ICG318 infusion.
  Renal Biopsies will be performed prior to and post-ICG318 infusion.
Complement levels | Assessed as per schedule of events up to 1 year after ICG318 infusion.
  Changes in C3 and C4 complement levels in serum.
Serum creatinine levels | Assessed as per schedule of events up to 1 year after ICG318 infusion.
Urine Protein-Creatinine Ratio (uPCR) levels. | Assessed as per schedule of events up to 1 year after ICG318 infusion.
eGFR value | Assessed as per schedule of events up to 1 year after ICG318 infusion.

IPD SHARING:
Plan to Share IPD: No